CLINICAL TRIAL: NCT03337373
Title: The Study of Pharmacokinetics and Pharmacodynamics of a Loading Dose Cisatracurium in Critically Ill Patients
Brief Title: The Study of Pharmacokinetics and Pharmacodynamics of Cisatracurium
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Panadda Panusitthikorn, Principal Investigator, Mahidol University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 06-60-07
Record Dates: First submitted 2017-11-02; First posted 2017-11-09 (Actual); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Critical Illness; Respiratory Distress Syndrome, Adult; Neuromuscular Blockade; Respiratory Failure; Paralysis; ARDS, Human
Keywords: Critical care; Neuromuscular Blocking Agents; Pharmacodynamics; Pharmacokinetics; Physiological Effects of Drugs
MeSH Terms: conditions — Critical Illness; Respiratory Distress Syndrome; Respiratory Insufficiency; Paralysis | interventions — cisatracurium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cisatracurium (Experimental): Patients who require paralysis with cisatracurium as part of their clinical care in ICU
  Interventions: Drug: cisatracurium

INTERVENTIONS:
Drug: cisatracurium — A single dose of 0.2 mg/kg intravenous bolus cisatracurium will be administered and blood samples will be taken before and at least 7 occasions post dose (at 1, 5, 10, 12, 15, 20, 30, and/or 60 minutes after a single bolus).
  Other Names: Nimbex

SUMMARY:
Pathophysiological changes influenced by multiple factors in critically ill patients, has a significant impact on pharmacokinetics (PK) and pharmacodynamics (PD) of cisatracurium. In order to understand better and find an appropriate dosing regimen, the purpose of this study is to investigate the PK and PD of a loading dose cisatracurium in critically ill patients.

Cisatracurium, nondepolarizing neuromuscular blocking agents (NMBAs), are commonly used in intensive care units because of a lesser effect on hemodynamic parameters and a reduction in mortality rate in ARDS patients. Loading dose recommended in clinical practice guidelines for sustained neuromuscular blockade in the adult critically ill patient is 0.1-0.2 mg/kg. Then, maintenance dose of 1-3 mcg/kg/min is followed regarding indications, such as ARDS. However, this recommended loading dose might not be adequate in critically ill patients, the study in this specific population might be needed.

DETAILED DESCRIPTION:
Neuromuscular blocking agents (NMBAs) are commonly used in critically ill patients, especially in adult respiratory distress syndrome (ARDS). Use of NMBAs to facilitate mechanical ventilation, to control patient/ventilator asynchrony and to reduce uncontrolled muscle tone in special conditions including tetanus, therapeutic hypothermia, and status epilepticus were increasingly found in current clinical practice.

Cisatracurium, 1Rcis-1'Rcis isomer of atracurium, is benzylisoquinolium nondepolarizing NMBAs which is three to five folds higher potency than atracurium besylate. The degradation of cisatracurium by hofmann elimination and ester hydrolysis in plasma generates laudanosine and a monoquaternary acrylate metabolite. Clinical practice guidelines for sustained neuromuscular blockade in the adult critically ill patient published in year 2016 strongly recommended cisatracurium due to a reduction in incidence of prolonged blockade, cardiovascular related adverse events and anaphylactic reactions. Moreover, recent evidence showed that early use of cisatracurium in early severe ARDS patients led to a significant reduction in mortality.

Regarding pharmacokinetics and pharmacodynamics of cisatracurium in critically ill patients, there were multiple factors affected cisatracurium blood concentration and neuromuscular blockade actions. Several reports demonstrated that pathophysiological changes, such as age, hypothermia/ hyperthermia, electrolyte imbalance and acid-base disturbances, had a significant impact on PK and PD of cisatracurium. Currently, there were an increasing data of slow response and less paralysis effect in critically ill patients receiving standard dose of cisatracurium. These may be explained by inadequate drug concentration at target organ, therefore, treatment failures regarding recommended dose of cisatracurium has been reported. Consequently, higher cisatracurium dose with higher drug concentration level might overcome a problem of inadequate level and therapeutic failure while receiving a standard dose of cisatracurium (a loading dose of 0.1-0.2 mg/kg, followed by a maintenance dose of 1-3 mcg/kg/min)

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years
* Admission for ICU care
* Require paralysis with cisatracurium as part of their clinical care
* Patients or legal representatives who are able to understand and are willing and able to give their signed informed consent before any trial-related procedures are performed

Exclusion Criteria:

* Lactating women
* Pregnancy women
* Documented history of hypersensitivity to cisatracurium
* Pre-existing neuromuscular disease
* Patients with burn lesions
* Currently diagnosed of hypothermia condition (tympanic body temperature ≤ 36 °C)
* Patients currently receiving intravenous bolus or push of cisatracurium within 24 hours or receiving intravenous continuous infusion of cisatracurium within 48 hours prior to enrollment
* Patients who have to receive intravenous continuous infusion of cisatracurium within 30 minutes after given intravenous bolus of 0.2 mg/ kg cisatracurium

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Total plasma concentration-time data | Pre-dose through 60 minutes post-dose
  Data will be collected in case-record form and managed by Microsoft Office Excel. Statistical analyses will be performed using SPSS.
Patient-ventilator asynchrony - time data | Pre-dose through 60 minutes post-dose
  Data will be collected in case-record form and managed by Microsoft Office Excel. Statistical analyses will be performed using SPSS.
The degree of neuromuscular block by train-of-four-watch monitor - time data | Pre-dose through 60 minutes post-dose
  Data will be collected in case-record form and managed by Microsoft Office Excel. Statistical analyses will be performed using SPSS.

SECONDARY OUTCOMES:
Time to maximum concentration | Pre-dose through 60 minutes post-dose
  Analysis of time to maximum concentration will be performed with a nonlinear mixed-effects population modelling approach as implemented in NONMEM software.
Half-life | Pre-dose through 60 minutes post-dose
  Analysis of half-life will be performed with a nonlinear mixed-effects population modelling approach as implemented in NONMEM software.
Clearance | Pre-dose through 60 minutes post-dose
  Analysis of clearance will be performed with a nonlinear mixed-effects population modelling approach as implemented in NONMEM software.
Elimination rate constant | Pre-dose through 60 minutes post-dose
  Analysis of elimination rate constant will be performed with a nonlinear mixed-effects population modelling approach as implemented in NONMEM software.
Time to maximum block | Pre-dose through 60 minutes post-dose
  Data will be collected in case-record form and managed by Microsoft Office Excel. Statistical analyses will be performed using SPSS.
Percentage of maximum block | Pre-dose through 60 minutes post-dose
  Data will be collected in case-record form and managed by Microsoft Office Excel. Statistical analyses will be performed using SPSS.
Time to patient-ventilator synchrony | Pre-dose through 60 minutes post-dose
  Data will be collected in case-record form and managed by Microsoft Office Excel. Statistical analyses will be performed using SPSS.

OTHER OUTCOMES:
Bispectral index (BIS) - time data | Pre-dose through 60 minutes post-dose
  Data will be collected in case-record form and managed by Microsoft Office Excel. Statistical analyses will be performed using SPSS.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Ramathibodi Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Liu X, Kruger PS, Weiss M, Roberts MS. The pharmacokinetics and pharmacodynamics of cisatracurium in critically ill patients with severe sepsis. Br J Clin Pharmacol. 2012 May;73(5):741-9. doi: 10.1111/j.1365-2125.2011.04149.x. PMID 22114771
- [Background] Murray MJ, DeBlock H, Erstad B, Gray A, Jacobi J, Jordan C, McGee W, McManus C, Meade M, Nix S, Patterson A, Sands MK, Pino R, Tescher A, Arbour R, Rochwerg B, Murray CF, Mehta S. Clinical Practice Guidelines for Sustained Neuromuscular Blockade in the Adult Critically Ill Patient. Crit Care Med. 2016 Nov;44(11):2079-2103. doi: 10.1097/CCM.0000000000002027. PMID 27755068
- [Background] Gainnier M, Roch A, Forel JM, Thirion X, Arnal JM, Donati S, Papazian L. Effect of neuromuscular blocking agents on gas exchange in patients presenting with acute respiratory distress syndrome. Crit Care Med. 2004 Jan;32(1):113-9. doi: 10.1097/01.CCM.0000104114.72614.BC. PMID 14707568
- [Background] Greenberg SB, Vender J. The use of neuromuscular blocking agents in the ICU: where are we now? Crit Care Med. 2013 May;41(5):1332-44. doi: 10.1097/CCM.0b013e31828ce07c. PMID 23591211
- [Background] Forel JM, Roch A, Marin V, Michelet P, Demory D, Blache JL, Perrin G, Gainnier M, Bongrand P, Papazian L. Neuromuscular blocking agents decrease inflammatory response in patients presenting with acute respiratory distress syndrome. Crit Care Med. 2006 Nov;34(11):2749-57. doi: 10.1097/01.CCM.0000239435.87433.0D. PMID 16932229
- [Background] Papazian L, Forel JM, Gacouin A, Penot-Ragon C, Perrin G, Loundou A, Jaber S, Arnal JM, Perez D, Seghboyan JM, Constantin JM, Courant P, Lefrant JY, Guerin C, Prat G, Morange S, Roch A; ACURASYS Study Investigators. Neuromuscular blockers in early acute respiratory distress syndrome. N Engl J Med. 2010 Sep 16;363(12):1107-16. doi: 10.1056/NEJMoa1005372. PMID 20843245
- [Background] Dieye E, Minville V, Asehnoune K, Conil C, Georges B, Cougot P, Fourcade O, Conil JM. Pharmacodynamics of cisatracurium in the intensive care unit: an observational study. Ann Intensive Care. 2014 Feb 11;4(1):3. doi: 10.1186/2110-5820-4-3. PMID 24521394
- [Background] Murray MJ, Cowen J, DeBlock H, Erstad B, Gray AW Jr, Tescher AN, McGee WT, Prielipp RC, Susla G, Jacobi J, Nasraway SA Jr, Lumb PD; Task Force of the American College of Critical Care Medicine (ACCM) of the Society of Critical Care Medicine (SCCM), American Society of Health-System Pharmacists, American College of Chest Physicians. Clinical practice guidelines for sustained neuromuscular blockade in the adult critically ill patient. Crit Care Med. 2002 Jan;30(1):142-56. doi: 10.1097/00003246-200201000-00021. No abstract available. PMID 11902255
- [Background] Welch RM, Brown A, Ravitch J, Dahl R. The in vitro degradation of cisatracurium, the R, cis-R'-isomer of atracurium, in human and rat plasma. Clin Pharmacol Ther. 1995 Aug;58(2):132-42. doi: 10.1016/0009-9236(95)90190-6. PMID 7648763
- [Background] McManus MC. Neuromuscular blockers in surgery and intensive care, Part 1. Am J Health Syst Pharm. 2001 Dec 1;58(23):2287-99. doi: 10.1093/ajhp/58.23.2287. PMID 11763807
- [Derived] Panusitthikorn P, Suthisisang C, Tangsujaritvijit V, Nosoongnoen W, Dilokpattanamongkol P. Pharmacokinetics and pharmacodynamics studies of a loading dose of cisatracurium in critically ill patients with respiratory failure. BMC Anesthesiol. 2022 Jan 22;22(1):32. doi: 10.1186/s12871-022-01571-2. PMID 35065599